CLINICAL TRIAL: NCT03441230
Title: ANTERO-AC-2: Determination of the Characteristics of Isometric Gastric Motility Measurement in Healthy Volunteers
Brief Title: Determination of the Characteristics of Isometric Gastric Motility Measurement in Healthy Volunteers
Acronym: ANTERO-AC-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Dr Jan Tack (Other)
Responsible Party: Sponsor-Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: S58817
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Gastroparesis
Keywords: stomach; motility
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Circumference of 13 cm, sphere form (diameter of 4 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 13 cm, cylinder form, length 11 cm (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 16 cm, sphere form (diameter of 5 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 16 cm, cylinder form, length 11 cm (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 16 cm, cylinder form, length 18 cm (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 19 cm, sphere form (diameter of 6 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 19 cm, cylinder form, length 11 cm (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 22 cm, sphere form (diameter of 7 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 25 cm, sphere form (diameter of 8 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics
- Circumference of 28 cm, sphere form (diameter of 9 cm) (Active Comparator)
  Interventions: Device: Balloon characteristics

INTERVENTIONS:
Device: Balloon characteristics — Different size balloon

SUMMARY:
There is a clear need for a novel method that can readily assess gastric motility in daily clinical practice. Isometric determination of the stomach motility would avoid the use of a large flaccid balloon while still being affordable. The aim of this study was to determine the optimal balloon characteristics that enable to measure motility-induced pressure changes in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* They are between 18-60 years old.
* Male and female.
* Patients must provide witnessed written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* They are older than 60 years old and younger than 18 years.
* They are taking medication.
* Have severely decreased kidney function.
* Have severely decreased liver function.
* Have severe heart disease, for example a history of irregular heartbeats, angina or heart attack.
* Have severe lung disease.
* Have severe psychiatric illness or neurological illness.
* Have any gastrointestinal disease.
* Have any dyspeptic symptoms.
* Women that are pregnant or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
Detection of distal stomach-induced contractions using various intragastric balloons | up to 1 year
  A comparison of various intragastric balloons for the assessment of gastric motility

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No